CLINICAL TRIAL: NCT06773819
Title: A Study on the Pathogenesis and Determinants of Intravenous Leiomyomatosis
Status: Not yet recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IVL001
Record Dates: First submitted 2024-12-30; First posted 2025-01-14 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Intravenous Leiomyomatosis; HPV Infection
Keywords: Intravenous leiomyomatosis; HPV
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Surgical specimen
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the impact of HPV infection in women with intravenous leiomyomatosis(IVL). The main question it aims to answer is:

Does HPV infection promote the development of IVL from uterine leiomyoma? Surgical sections and HPV-DNA test results will be collected in participants diagnosed with IVL or uterine leiomyoma.

DETAILED DESCRIPTION:
Previous proteomic studies have demonstrated that HPV infection-related proteins are more highly expressed in intravenous leiomyomatosis (IVL) compared to uterine leiomyoma (uML). Consequently, we conducted a case-control study to investigate the association between HPV and the development of IVL. We recruited adult patients diagnosed with either IVL or uML, collected their medical histories, surgical specimens from various sites, and HPV-DNA test results from cervical exfoliated cells, and performed subsequent statistical analyses and mechanistic investigations.

ELIGIBILITY:
Inclusion Criteria:

* Adult female patients with suspected IVL or uterine leiomyoma who receive surgery at PUMCH
* Be able to understand and sign the informed consent

Exclusion Criteria:

* Patients with other concurrent malignant tumors
* Pregnant or lactating female
* Postoperative pathology do not include IVL or uterine leiomyoma

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Adult female patients with suspected IVL
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
HPV-DNA test result | From date of enrollment until the date of surgery at PUMCH or date of death from any cause, whichever came first, assessed up to 100 months

IPD SHARING:
Plan to Share IPD: Undecided